CLINICAL TRIAL: NCT00272883
Title: Molecular Analysis of Neuromuscular Disease
Brief Title: Molecular and Genetic Studies of Congenital Myopathies
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Alan H. Beggs, Sir Edwin & Lady Manton Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: 03-08-128R; AR44345; NS40828
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Central Core Disease; Centronuclear Myopathy; Congenital Fiber Type Disproportion; Multiminicore Disease; Myotubular Myopathy; Nemaline Myopathy; Rigid Spine Muscular Dystrophy; Undefined Congenital Myopathy
Keywords: central core; centronuclear; multiminicore; multicore; minicore; congenital fiber type disproportion; myotubular; nemaline; congenital myopathy; neuromuscular; rigid spine
MeSH Terms: conditions — Myopathy, Central Core; Myopathies, Structural, Congenital; Minicore Myopathy with External Ophthalmoplegia; Myopathies, Nemaline; Myotonia Congenita

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The primary biospecimens retained are blood, saliva and muscle tissue samples. Other specimens are retained on a case-by-case basis.
Oversight: Data Monitoring Committee: No

SUMMARY:
In the Congenital Myopathy Research Program at Boston Children's Hospital and Harvard Medical School, the researchers are studying the congenital myopathies (neuromuscular diseases present from birth), including central core disease, centronuclear/myotubular myopathy, congenital fiber type disproportion, multiminicore disease, nemaline myopathy, rigid spine muscular dystrophy, SELENON (SEPN1), RYR1 myopathy, ADSS1 (ADSSL) Myopathy and undefined congenital myopathies. The primary goal of the research is to better understand the genes and proteins (gene products) involved in muscle functioning and disease. The researchers hope that our studies will allow for improved diagnosis and treatment of individuals with congenital myopathies in the future. For more information, visit the Laboratory Website at www.childrenshospital.org/research/beggs

DETAILED DESCRIPTION:
The Congenital Myopathy Research Program consists of a group of scientists and healthcare providers all working to better understand the congenital myopathies. We are taking two approaches to reach our research goals. The first involves identifying and describing new genes and proteins involved in the skeletal muscles that allow our bodies to move. Simultaneously, studies are underway to identify genetic changes (mutations) that cause human neuromuscular disease. Thus, our second approach is to identify mutations, learn how they are inherited in families, and understand how they lead to weakness in individuals with neuromuscular disease. These approaches allow correlation of our basic muscle biology findings with our studies on muscle tissue of affected individuals.

Our research would not be possible without the generous participation of individuals and families with congenital myopathies. Participation in our studies is free of charge. Travel to Boston is not required, and we welcome the participation of individuals from around the world.

We appreciate the participation of all individuals with a congenital myopathy, as well as their first-degree relatives. Participants with a congenital myopathy are asked to donate medical records, a blood or saliva sample, and a muscle tissue sample (if available). Participating relatives are asked to donate a blood sample. The blood/saliva sample is used to acquire DNA (genetic material) which can be used to identify genetic changes and to study how a disease is inherited in a family. The medical records are employed to understand a participant's symptoms. The muscle tissue is used to better understand the disease at the muscular level by studying the gene expression and protein levels in individuals with congenital myopathies.

For more information, visit the Laboratory Website at www.childrenshospital.org/research/beggs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a clinical or suspected diagnosis of a congenital myopathy and their family members

Exclusion Criteria:

* No specific exclusion criteria. Our studies do not include myotonia congenita or related conditions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a clinical or suspected diagnosis of a congenital myopathy and their family members.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2003-08; Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Identification of Neuromuscular Disease Genes | The time frame for disease gene discovery is unpredictable and may range from several days to several decades.
  This is an ongoing genetic discovery study aimed at finding and confirming pathogenic mutations in known and new disease genes.

SECONDARY OUTCOMES:
Characterization of Clinical Features of Congenital Myopathies | The time frame for disease classification and genotype-phenotype correlation is unpredictable and may range from several days to several decades.
  As known as known and new disease genes are identified the resulting genotypes are correlated with subject phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Alan H. Beggs, Ph.D., Principal Investigator — Children's Hospital Boston/Harvard Medical School
Locations (1):
- Genetics Division, Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Pierson CR, Tomczak K, Agrawal P, Moghadaszadeh B, Beggs AH. X-linked myotubular and centronuclear myopathies. J Neuropathol Exp Neurol. 2005 Jul;64(7):555-64. doi: 10.1097/01.jnen.0000171653.17213.2e. PMID 16042307
- [Result] Agrawal PB, Strickland CD, Midgett C, Morales A, Newburger DE, Poulos MA, Tomczak KK, Ryan MM, Iannaccone ST, Crawford TO, Laing NG, Beggs AH. Heterogeneity of nemaline myopathy cases with skeletal muscle alpha-actin gene mutations. Ann Neurol. 2004 Jul;56(1):86-96. doi: 10.1002/ana.20157. PMID 15236405
- [Result] Ryan MM, Ilkovski B, Strickland CD, Schnell C, Sanoudou D, Midgett C, Houston R, Muirhead D, Dennett X, Shield LK, De Girolami U, Iannaccone ST, Laing NG, North KN, Beggs AH. Clinical course correlates poorly with muscle pathology in nemaline myopathy. Neurology. 2003 Feb 25;60(4):665-73. doi: 10.1212/01.wnl.0000046585.81304.bc. PMID 12601110
- [Result] Ryan MM, Schnell C, Strickland CD, Shield LK, Morgan G, Iannaccone ST, Laing NG, Beggs AH, North KN. Nemaline myopathy: a clinical study of 143 cases. Ann Neurol. 2001 Sep;50(3):312-20. doi: 10.1002/ana.1080. PMID 11558787
- [Result] Sanoudou D, Frieden LA, Haslett JN, Kho AT, Greenberg SA, Kohane IS, Kunkel LM, Beggs AH. Molecular classification of nemaline myopathies: "nontyping" specimens exhibit unique patterns of gene expression. Neurobiol Dis. 2004 Apr;15(3):590-600. doi: 10.1016/j.nbd.2003.12.013. PMID 15056467
- [Result] Sanoudou D, Haslett JN, Kho AT, Guo S, Gazda HT, Greenberg SA, Lidov HG, Kohane IS, Kunkel LM, Beggs AH. Expression profiling reveals altered satellite cell numbers and glycolytic enzyme transcription in nemaline myopathy muscle. Proc Natl Acad Sci U S A. 2003 Apr 15;100(8):4666-71. doi: 10.1073/pnas.0330960100. Epub 2003 Apr 3. PMID 12677001
- [Result] Wattanasirichaigoon D, Swoboda KJ, Takada F, Tong HQ, Lip V, Iannaccone ST, Wallgren-Pettersson C, Laing NG, Beggs AH. Mutations of the slow muscle alpha-tropomyosin gene, TPM3, are a rare cause of nemaline myopathy. Neurology. 2002 Aug 27;59(4):613-7. doi: 10.1212/wnl.59.4.613. PMID 12196661
- [Result] Nowak KJ, Wattanasirichaigoon D, Goebel HH, Wilce M, Pelin K, Donner K, Jacob RL, Hubner C, Oexle K, Anderson JR, Verity CM, North KN, Iannaccone ST, Muller CR, Nurnberg P, Muntoni F, Sewry C, Hughes I, Sutphen R, Lacson AG, Swoboda KJ, Vigneron J, Wallgren-Pettersson C, Beggs AH, Laing NG. Mutations in the skeletal muscle alpha-actin gene in patients with actin myopathy and nemaline myopathy. Nat Genet. 1999 Oct;23(2):208-12. doi: 10.1038/13837. PMID 10508519
- [Result] North KN, Yang N, Wattanasirichaigoon D, Mills M, Easteal S, Beggs AH. A common nonsense mutation results in alpha-actinin-3 deficiency in the general population. Nat Genet. 1999 Apr;21(4):353-4. doi: 10.1038/7675. No abstract available. PMID 10192379
- [Result] Pelin K, Hilpela P, Donner K, Sewry C, Akkari PA, Wilton SD, Wattanasirichaigoon D, Bang ML, Centner T, Hanefeld F, Odent S, Fardeau M, Urtizberea JA, Muntoni F, Dubowitz V, Beggs AH, Laing NG, Labeit S, de la Chapelle A, Wallgren-Pettersson C. Mutations in the nebulin gene associated with autosomal recessive nemaline myopathy. Proc Natl Acad Sci U S A. 1999 Mar 2;96(5):2305-10. doi: 10.1073/pnas.96.5.2305. PMID 10051637
- [Result] Ottenheijm CA, Lawlor MW, Stienen GJ, Granzier H, Beggs AH. Changes in cross-bridge cycling underlie muscle weakness in patients with tropomyosin 3-based myopathy. Hum Mol Genet. 2011 May 15;20(10):2015-25. doi: 10.1093/hmg/ddr084. Epub 2011 Feb 28. PMID 21357678
- [Result] Lawlor MW, Dechene ET, Roumm E, Geggel AS, Moghadaszadeh B, Beggs AH. Mutations of tropomyosin 3 (TPM3) are common and associated with type 1 myofiber hypotrophy in congenital fiber type disproportion. Hum Mutat. 2010 Feb;31(2):176-83. doi: 10.1002/humu.21157. PMID 19953533
- [Result] Ottenheijm CA, Hooijman P, DeChene ET, Stienen GJ, Beggs AH, Granzier H. Altered myofilament function depresses force generation in patients with nebulin-based nemaline myopathy (NEM2). J Struct Biol. 2010 May;170(2):334-43. doi: 10.1016/j.jsb.2009.11.013. Epub 2009 Nov 26. PMID 19944167
- [Result] Laing NG, Dye DE, Wallgren-Pettersson C, Richard G, Monnier N, Lillis S, Winder TL, Lochmuller H, Graziano C, Mitrani-Rosenbaum S, Twomey D, Sparrow JC, Beggs AH, Nowak KJ. Mutations and polymorphisms of the skeletal muscle alpha-actin gene (ACTA1). Hum Mutat. 2009 Sep;30(9):1267-77. doi: 10.1002/humu.21059. PMID 19562689
- [Result] Ottenheijm CA, Witt CC, Stienen GJ, Labeit S, Beggs AH, Granzier H. Thin filament length dysregulation contributes to muscle weakness in nemaline myopathy patients with nebulin deficiency. Hum Mol Genet. 2009 Jul 1;18(13):2359-69. doi: 10.1093/hmg/ddp168. Epub 2009 Apr 4. PMID 19346529
- [Result] Lehtokari VL, Greenleaf RS, DeChene ET, Kellinsalmi M, Pelin K, Laing NG, Beggs AH, Wallgren-Pettersson C. The exon 55 deletion in the nebulin gene--one single founder mutation with world-wide occurrence. Neuromuscul Disord. 2009 Mar;19(3):179-81. doi: 10.1016/j.nmd.2008.12.001. Epub 2009 Feb 15. PMID 19232495
- [Result] Pierson CR, Agrawal PB, Blasko J, Beggs AH. Myofiber size correlates with MTM1 mutation type and outcome in X-linked myotubular myopathy. Neuromuscul Disord. 2007 Jul;17(7):562-8. doi: 10.1016/j.nmd.2007.03.010. Epub 2007 May 29. PMID 17537630
- [Result] Agrawal PB, Greenleaf RS, Tomczak KK, Lehtokari VL, Wallgren-Pettersson C, Wallefeld W, Laing NG, Darras BT, Maciver SK, Dormitzer PR, Beggs AH. Nemaline myopathy with minicores caused by mutation of the CFL2 gene encoding the skeletal muscle actin-binding protein, cofilin-2. Am J Hum Genet. 2007 Jan;80(1):162-7. doi: 10.1086/510402. Epub 2006 Nov 14. PMID 17160903
- See also: The Beggs lab website — http://www.childrenshospital.org/research/beggs